CLINICAL TRIAL: NCT02947633
Title: Sciatic Peripheral Nerve Blockade for Pain Control Following Hamstring Autograft Harvest in Adolescents: A Comparison of Two Techniques
Brief Title: Sciatic Technique Comparison of Nerve Blockade for Pain Control Following Hamstring Autograft Harvest in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-6533
Record Dates: First submitted 2015-11-11; First posted 2016-10-28 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament (ACL) Tear
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous sciatic PNB (Experimental): If a CPI catheter is placed, the CPI catheter will be placed under ultra-sound guidance, with the tip of the catheter being placed immediately adjacent to the sciatic nerve, after the local anesthesia has been deposited. CPI catheters will only remain in-situ for 48 hours.
  Interventions: Drug: Continuous sciatic PNB
- Single-injection sciatic PNB (Active Comparator): Under ultrasound-guidance, the sciatic nerve can readily be identified in the posterior thigh. The nerve appears hyperechoic and can be traced distally to the popliteal fossa, where it divides into the tibial and common peroneal nerves. Local anesthesia is injected under real-time visualization following a negative aspiration. If a single-injection block is done, local anesthesia is deposited adjacent to the sciatic nerve within the fascial plane, but not within the epineurium. As such, single-injection sciatic PNB, which can last up to 24 hours, should provide adequate analgesia precluding the need for oral narcotic or nonsteroidal anti-inflammatory medications following ACL reconstruction with a hamstring autograft.
  Interventions: Drug: Single-injection sciatic PNB

INTERVENTIONS:
Drug: Single-injection sciatic PNB — Single-injection sciatic PNB is a regional anesthetic technique employed to anesthetize the sciatic nerve with a single dose of local anesthetic. This technique offers pain control for a limited amount of time based on the volume and concentration of local anesthetic used.
  Arms: Single-injection sciatic PNB
Drug: Continuous sciatic PNB — Continuous sciatic PNB entails placing a continuous perineural infusion (CPI) catheter so that local anesthetic may be released slowly but continuously adjacent to the sciatic nerve (perineural) for several days postoperatively. The continuous PNB has the ability to reliably provide analgesia on subsequent postoperative days.
  Participants my be randomized to receive an additional experimental continuous pain ball during surgery which can provide up to 48 hours of pain relief.
  Arms: Continuous sciatic PNB

SUMMARY:
The purpose of this research is to compare the effect of single-injection sciatic PNB to continuous sciatic PNB on 1) postoperative pain control as measured by self-reported pain scores, pain medication use, and unplanned hospital admission due to poor pain control, 2) active knee flexion, and 3) patient satisfaction with pain control following ACL reconstruction with a hamstring autograft. The results of this research have the potential to positively impact pain control for the adolescent population undergoing this surgical procedure and foster responsible utilization of limited resources.

DETAILED DESCRIPTION:
SPECIFIC AIM 1. The first aim of the study is to explore the impact of sciatic PNB technique on hamstring donor site pain control postoperatively.

H1.a. The extended duration of analgesia offered by continuous sciatic PNB decreases pain scores during the initial 72 hours following hamstring autograft harvest when compared to single-injection sciatic PNB.

H1.b. The extended duration of analgesia offered by continuous sciatic PNB decreases oral pain medication use during the initial 72 hours following hamstring autograft harvest when compared to single-injection sciatic PNB.

H1.c. The extended duration of analgesia offered by continuous sciatic PNB decreases the incidence of unplanned admission due to poor pain control during the initial 72 hours following hamstring autograft harvest when compared to single-injection sciatic PNB.

SPECIFIC AIM 2. The second aim of the study is to explore the impact of sciatic PNB technique on active knee flexion postoperatively.

H2. The extended duration of analgesia offered by continuous sciatic PNB does not delay active knee flexion during the initial 72 hours following hamstring autograft harvest when compared to single-injection sciatic PNB.

SPECIFIC AIM 3. The third aim of the study is to explore the impact of sciatic PNB technique on patient satisfaction with postoperative pain control.

H3.1. The extended duration of analgesia offered by continuous sciatic PNB improves patient satisfaction during the initial 72 hours following hamstring autograft harvest when compared to single-injection sciatic PNB.

ELIGIBILITY:
Inclusion Criteria:

A subject may be INCLUDED in this study if:

1. The subject is male or female;
2. The subject is of any racial or ethnic group;
3. The subject is age 10 years to 18 years (inclusive);
4. The subject is scheduled for the following: Unilateral ACL reconstruction with a hamstring autograft under general anesthesia on an outpatient basis, and not being performed in conjunction with any other surgical procedures;
5. The subject is American Society of Anesthesiologists (ASA) patient classification I-II;
6. The subject or legally authorized representative has consented to femoral and sciatic peripheral nerve blockade for the procedure and the consent for peripheral nerve blockade has been obtained by a clinician (MD, DO, CRNA or APN) authorized to obtain consent;
7. The subject's legally authorized representative has given written informed consent to participate in the study and when appropriate, the subject has given assent or consent to participate.

Exclusion Criteria:

A subject will be EXCLUDED from this study if:

1. Additional surgical procedures are being performed concurrently;
2. The subject is ASA classification > II;
3. The subject has pre-existing allergies to amide local anesthetics;
4. The subject receives sedation preoperatively;
5. The subject is schedule for overnight hospital admission;
6. The subject has any other condition, which in the opinion of the principal investigator, would not be suitable for participation in the study, including but not limited to coagulopathy, preexisting central or peripheral nervous systems disorders, and local infection or sores at the anticipated site of needle insertion;
7. Unsuccessful PNB or CPI catheter placement occurs during the study. -

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Pain Reduction | 72 Hours
  Guardian collects pain data for 72 hours post ACL through self-reported pain scores.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Furstein, CRNA, Principal Investigator — AANA Foundation
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agin CW, Glass PSA. Tolerance and aging: optimizing analgesia in pain management. Anesth Analg. 2005 Jun;100(6):1731-1732. doi: 10.1213/01.ANE.0000152203.17541.16. No abstract available. PMID 15920205
- [Background] Beales JG, Holt PJ, Keen JH, Mellor VP. Children with juvenile chronic arthritis: their beliefs about their illness and therapy. Ann Rheum Dis. 1983 Oct;42(5):481-6. doi: 10.1136/ard.42.5.481. PMID 6625698
- [Background] Bushnell BD, Sakryd G, Noonan TJ. Hamstring donor-site block: evaluation of pain control after anterior cruciate ligament reconstruction. Arthroscopy. 2010 Jul;26(7):894-900. doi: 10.1016/j.arthro.2009.11.022. Epub 2010 May 13. PMID 20620788
- [Background] Distad BJ, Weiss MD. Clinical and electrodiagnostic features of sciatic neuropathies. Phys Med Rehabil Clin N Am. 2013 Feb;24(1):107-20. doi: 10.1016/j.pmr.2012.08.023. Epub 2012 Oct 31. PMID 23177034
- [Background] Frost S, Grossfeld S, Kirkley A, Litchfield B, Fowler P, Amendola A. The efficacy of femoral nerve block in pain reduction for outpatient hamstring anterior cruciate ligament reconstruction: a double-blind, prospective, randomized trial. Arthroscopy. 2000 Apr;16(3):243-8. doi: 10.1016/s0749-8063(00)90047-1. PMID 10750003
- [Background] Gagnier JJ, Morgenstern H, Chess L. Interventions designed to prevent anterior cruciate ligament injuries in adolescents and adults: a systematic review and meta-analysis. Am J Sports Med. 2013 Aug;41(8):1952-62. doi: 10.1177/0363546512458227. Epub 2012 Sep 12. PMID 22972854
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Mathews L. Pain in children: neglected, unaddressed and mismanaged. Indian J Palliat Care. 2011 Jan;17(Suppl):S70-3. doi: 10.4103/0973-1075.76247. PMID 21811376
- [Background] Mehta VM, Mandala C, Foster D, Petsche TS. Comparison of revision rates in bone-patella tendon-bone autograft and allograft anterior cruciate ligament reconstruction. Orthopedics. 2010 Jan;33(1):12. doi: 10.3928/01477447-20091124-15. PMID 20055340
- [Background] Pallis M, Svoboda SJ, Cameron KL, Owens BD. Survival comparison of allograft and autograft anterior cruciate ligament reconstruction at the United States Military Academy. Am J Sports Med. 2012 Jun;40(6):1242-6. doi: 10.1177/0363546512443945. Epub 2012 Apr 24. PMID 22534281
- [Background] Pinczewski LA, Lyman J, Salmon LJ, Russell VJ, Roe J, Linklater J. A 10-year comparison of anterior cruciate ligament reconstructions with hamstring tendon and patellar tendon autograft: a controlled, prospective trial. Am J Sports Med. 2007 Apr;35(4):564-74. doi: 10.1177/0363546506296042. Epub 2007 Jan 29. PMID 17261567
- [Background] Shaw T, Williams MT, Chipchase LS. Do early quadriceps exercises affect the outcome of ACL reconstruction? A randomised controlled trial. Aust J Physiother. 2005;51(1):9-17. doi: 10.1016/s0004-9514(05)70048-9. PMID 15748120
- [Background] Silvers HJ, Mandelbaum BR. Prevention of anterior cruciate ligament injury in the female athlete. Br J Sports Med. 2007 Aug;41 Suppl 1(Suppl 1):i52-9. doi: 10.1136/bjsm.2007.037200. Epub 2007 Jul 3. PMID 17609222
- [Background] Tran KM, Ganley TJ, Wells L, Ganesh A, Minger KI, Cucchiaro G. Intraarticular bupivacaine-clonidine-morphine versus femoral-sciatic nerve block in pediatric patients undergoing anterior cruciate ligament reconstruction. Anesth Analg. 2005 Nov;101(5):1304-1310. doi: 10.1213/01.ANE.0000180218.54037.0B. PMID 16243985
- [Background] Twycross A. Educating nurses about pain management: the way forward. J Clin Nurs. 2002 Nov;11(6):705-14. doi: 10.1046/j.1365-2702.2002.00677.x. PMID 12427174
- [Background] Wegener JT, van Ooij B, van Dijk CN, Hollmann MW, Preckel B, Stevens MF. Value of single-injection or continuous sciatic nerve block in addition to a continuous femoral nerve block in patients undergoing total knee arthroplasty: a prospective, randomized, controlled trial. Reg Anesth Pain Med. 2011 Sep-Oct;36(5):481-8. doi: 10.1097/AAP.0b013e318228c33a. PMID 21857273
- [Background] Kimberlin CL, Winterstein AG. Validity and reliability of measurement instruments used in research. Am J Health Syst Pharm. 2008 Dec 1;65(23):2276-84. doi: 10.2146/ajhp070364. PMID 19020196